CLINICAL TRIAL: NCT00027625
Title: A Phase I Study Of ZD 1839 And Temozolomide For The Treatment Of Gliomas
Brief Title: Gefitinib Plus Temozolomide in Treating Patients With Malignant Primary Glioma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: NABTC-0102; CDR0000069049 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2001-12-07; First posted 2003-01-27 (Estimated); Last update posted 2018-06-27 (Actual); Status verified 2018-06

CONDITIONS: Brain and Central Nervous System Tumors
Keywords: recurrent adult brain tumor; adult glioblastoma; adult anaplastic astrocytoma; adult anaplastic oligodendroglioma; adult mixed glioma; adult giant cell glioblastoma; adult gliosarcoma
MeSH Terms: conditions — Central Nervous System Neoplasms; Brain Neoplasms; Glioblastoma; Astrocytoma; Oligodendroglioma; Glioma; Gliosarcoma | interventions — Gefitinib; Temozolomide

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

INTERVENTIONS:
Drug: gefitinib
Drug: temozolomide

SUMMARY:
RATIONALE: Biological therapies such as gefitinib may interfere with the growth of cancer cells and slow the growth of the tumor. Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining gefitinib with chemotherapy may kill more tumor cells.

PURPOSE: Phase I trial to study the effectiveness of combining gefitinib with temozolomide in treating patients who have malignant primary glioma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the maximum tolerated dose of gefitinib when given in combination with temozolomide in patients with malignant primary glioma.
* Determine the toxic effects of this regimen in these patients.
* Determine the pharmacokinetics of this regimen in these patients.

OUTLINE: This is a multicenter, dose-escalation study of gefitinib. Patients are stratified according to use of concurrent enzyme-inducing anti-epileptic drugs (yes vs no).

Patients receive oral gefitinib once daily on days 1-35 and oral temozolomide once daily on days 8-12 for the first course only. For the second and subsequent courses, patients receive oral gefitinib once daily on days 1-28 and oral temozolomide once daily on days 1-5. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-6 patients receive escalating doses of gefitinib until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity.

Patients are followed every 2 months for 1 year and then every 3-6 months thereafter.

PROJECTED ACCRUAL: Approximately 3-42 patients will be accrued for this study within 1-14 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed malignant primary glioma

  * Glioblastoma multiforme
  * Anaplastic astrocytoma
  * Anaplastic oligodendroglioma
  * Anaplastic mixed oligoastrocytoma
  * Malignant astrocytoma not otherwise specified
* Stable or progressive disease

  * Progressive disease after interstitial brachytherapy or stereotactic radiosurgery must be confirmed by positron emission tomography or thallium scan, magnetic resonance spectroscopy, or surgical biopsy
* Prior treatment for no more than 3 prior relapses allowed

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* Karnofsky 60-100%

Life expectancy:

* More than 8 weeks

Hematopoietic:

* WBC greater than 3,000/mm^3
* Absolute neutrophil count greater than 1,500/mm^3
* Platelet count greater than 120,000/mm^3
* Hemoglobin greater than 10 g/dL (transfusion allowed)

Hepatic:

* Bilirubin less than 1.5 times upper limit of normal (ULN)
* SGOT less than 1.5 times ULN

Renal:

* Creatinine less than 1.5 mg/dL OR
* Creatinine clearance greater than 60 mL/min

Other:

* Not pregnant
* Negative pregnancy test
* Fertile patients must use effective contraception
* No active infection
* No other concurrent significant medical illness that would preclude study participation
* No significant gastrointestinal risk factors (e.g., active ulcerative colitis) within the past 6 months
* No other malignancy within the past 3 years except non-melanoma skin cancer or carcinoma in situ of the cervix

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* At least 1 week since prior interferon
* No concurrent filgrastim (G-CSF) during the first course of study therapy

Chemotherapy:

* At least 2 weeks since prior vincristine
* At least 3 weeks since prior procarbazine
* At least 6 weeks since prior nitrosoureas
* Prior or concurrent temozolomide allowed if there is no evidence of progression while receiving therapy

Endocrine therapy:

* At least 1 week since prior tamoxifen
* Must be on a stable dose of corticosteroids for at least 5 days

Radiotherapy:

* See Disease Characteristics
* At least 3 weeks since prior radiotherapy

Surgery:

* See Disease Characteristics
* At least 1 week since prior surgical resection

Other:

* Recovered from all prior therapy
* No prior gefitinib
* At least 1 week since prior non-cytotoxic agents except radiosensitizers
* At least 4 weeks since prior cytotoxic therapy
* At least 4 weeks since prior investigational agents
* At least 3 years since prior therapy for other malignancy
* Concurrent therapeutic agents allowed at stable dosage
* Concurrent enzyme-inducing anti-epileptic drugs allowed if continued during study participation

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2002-01-28 (Actual); Primary Completion 2005-03-17 (Actual); Study Completion 2005-11-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Prados, MD, Study Chair — UCSF Medical Center at Parnassus
Locations (11):
- United States (11):
  - Jonsson Comprehensive Cancer Center, UCLA, Los Angeles, California
  - UCSF Comprehensive Cancer Center, San Francisco, California
  - Warren Grant Magnuson Clinical Center - NCI Clinical Studies Support, Bethesda, Maryland
  - Dana-Farber/Harvard Cancer Center at Dana Farber Cancer Institute, Boston, Massachusetts
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - University of Pittsburgh Cancer Institute, Pittsburgh, Pennsylvania
  - Simmons Cancer Center - Dallas, Dallas, Texas
  - University of Texas - MD Anderson Cancer Center, Houston, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - University of Wisconsin Comprehensive Cancer Center, Madison, Wisconsin

REFERENCES:
- [Result] Prados MD, Yung WK, Wen PY, Junck L, Cloughesy T, Fink K, Chang S, Robins HI, Dancey J, Kuhn J. Phase-1 trial of gefitinib and temozolomide in patients with malignant glioma: a North American brain tumor consortium study. Cancer Chemother Pharmacol. 2008 May;61(6):1059-67. doi: 10.1007/s00280-007-0556-y. Epub 2007 Aug 11. PMID 17694310